CLINICAL TRIAL: NCT00791479
Title: Assessment of Dose-Dependent Effects of LY2189265 on Glycemic Control in Patients With Type 2 Diabetes Treated Only With Lifestyle Interventions
Brief Title: Effects of LY2189265 on Glycemic Control in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12565; H9X-MC-GBCK (Other: Eli Lilly and Company); CTRI/2009/091/000105 (Registry Identifier: India)
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes, type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 0.1 milligram (mg) LY2189265 (Experimental): LY2189265: 0.1 milligram (mg), subcutaneous (SC), once weekly (QW)
  Interventions: Drug: LY2189265 and Lifestyle Measures
- 0.5 milligram (mg) LY2189265 (Experimental): LY2189265: 0.5 milligram (mg), subcutaneous (SC), once weekly (QW)
  Interventions: Drug: LY2189265 and Lifestyle Measures
- 1.0 milligram (mg) LY2189265 (Experimental): LY2189265: 1.0 milligram (mg), subcutaneous (SC), once weekly (QW)
  Interventions: Drug: LY2189265 and Lifestyle Measures
- 1.5 milligram (mg) LY2189265 (Experimental): LY2189265: 1.5 milligram (mg), subcutaneous (SC), once weekly (QW)
  Interventions: Drug: LY2189265 and Lifestyle Measures
- Placebo (Placebo Comparator): Placebo: subcutaneous (SC) once weekly (QW)
  Interventions: Drug: Placebo solution and Lifestyle Measures

INTERVENTIONS:
Drug: LY2189265 and Lifestyle Measures — Subcutaneous injection once-weekly for up to 12 weeks
  Other Names: Dulaglutide
  Arms: 0.1 milligram (mg) LY2189265; 0.5 milligram (mg) LY2189265; 1.0 milligram (mg) LY2189265; 1.5 milligram (mg) LY2189265
Drug: Placebo solution and Lifestyle Measures — Subcutaneous injection once-weekly for up to 12 weeks
  Arms: Placebo

SUMMARY:
This is a study to demonstrate that different doses of once-weekly LY2189265 injected subcutaneously will have dose proportional effect on hemoglobin A1c (HbA1c) at 12 weeks in participants with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Participants in the trial will be randomized to one of the LY2189265 doses (4 doses are planned, range 0.1-1.5 milligram [mg]) or placebo. The main purpose is to assess dose-dependent effect of this new compound on blood glucose over a period of 12 weeks. Therefore, glycosylated hemoglobin (HbA1c) is chosen as the primary efficacy measure. Several other attributes of glycemic control and endocrine function of pancreas will be assessed as secondary objectives. These secondary objectives will be used to compare the effect of the experimental compound and placebo. Since LY2189265 is in early phase of development, comprehensive safety assessment is planned to learn more about possible side-effects and to establish benefit/risk profile of individual doses of the drug. The trial is organized in four phases: screening, lead-in period to establish baseline status of participants in each group, treatment period during which participants will be randomized into 1 of 5 groups (4 will receive one of the LY2189265 doses, 1 group will receive placebo), and safety follow up. Maximum of 9 study visits are planned. Study drug (LY2189265 or placebo) will be administered once weekly via subcutaneous (SC) injections. Rescue intervention was allowed after randomization for those participants whose hyperglycemia reached pre-defined unacceptable high values. Participants on rescue therapy remained in the study and continued to receive study drug. Participants who received rescue therapy were included in the analysis population, but only measurements obtained prior to the beginning of rescue therapy were included in specified efficacy analyses.

A 3-mg LY2189265 dose was discontinued and replaced with the 1.5 mg dose based on dose finding Study H9X-MC-GBCF; NCT00734474. Except where noted, data summaries from the 3 discontinued 3-mg LY2189265 participants (n=3) are not included due to the small number of participants and the short treatment duration.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, type 2
* Treatment regimens: diet and exercise only or are taking metformin as monotherapy and are willing to discontinue this medication
* Have completed at least 8 weeks of wash-out prior to randomization (if on metformin therapy at screening)
* Have a qualifying glycosylated hemoglobin (HbA1c) value, as determined by the central laboratory: at screening (for diet and exercise only ≥7.0% to ≤9.5%; for metformin monotherapy >6.5% to ≤9.0%) and at time of randomization for all participants ≥6.5% to ≤9.5%
* Females of childbearing potential must test negative for pregnancy and agree to use a reliable birth control method
* Have a body mass index (BMI) between 23 and 40 kilograms/meter squared (kg/m^2), inclusive, for participants who are native to, and reside in, South and/or East Asia; all other participants must have a BMI between 25 and 40 kg/m^2, inclusive.
* Stable weight for 3 months prior to screening

Exclusion Criteria:

* Diabetes mellitus, type 1
* Taking any glucose-lowering oral agents other than metformin within 3 months prior to screening
* Use of glucagon-like peptide-1 (GLP-1) analog (for example, exenatide) within 6 months prior to screening or being treated within insulin (with the exception of short-term management of acute conditions that occurred more than 3 months immediately prior to screening)
* Use of medications (prescription or over-the counter) to promote weight loss
* Chronic (>2 weeks) use of systemic glucocorticoid therapy
* Gastric emptying abnormality, history of bariatric surgery or chronic use of drugs that affect gastrointestinal motility
* Use of central nervous system (CNS) stimulant (for example, Ritalin-sustained release [SR])
* Cardiovascular event within 6 months prior to screening
* Poorly controlled hypertension (determined by a mean seated systolic blood pressure (BP) ≥160 millimeters of mercury (mmHg) or mean seated diastolic BP ≥95 mmHg at screening or randomization)
* Electrocardiogram (ECG) reading considered outside the normal limits by the investigator and relevant for interpretation or indicating cardiac disease
* Liver disease, hepatitis, chronic hepatitis, or alanine transaminase levels >3.0 times upper limit of normal
* Clinical signs or symptoms of pancreatitis or history of chronic or acute pancreatitis at time of screening
* Amylase ≥3 times the upper limit of normal and/or lipase ≥2 times upper limit of normal which are determined by central labs at the time of screening
* Serum creatinine ≥1.5 milligrams per deciliter (mg/dL) for men or ≥1.4 mg/dL for women or a creatinine clearance <60 milliliter (mL)/minute which are determined by central labs at the time of screening
* Uncontrolled diabetes (defined as 2 or more episode of hyperosmolar state requiring hospitalization in the 6 months prior to screening)
* Significant active, uncontrolled endocrine or autoimmune abnormality
* History of a transplanted organ (corneal transplants are allowed)
* Active or untreated malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years
* Have any other condition, in the opinion of the investigator, that may preclude the participant from following or completing the protocol
* Investigator site personnel directly affiliated with this study and/or their immediate families (spouse, parent, child, or sibling, whether biological or legally adopted)
* Sponsor employees
* Received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Participated in an interventional medical, surgical, or pharmaceutical study within 30 days prior to entry into the study
* Have previously completed or withdrawn from this study after providing informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (45):
- United States (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Springs, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vincennes, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomfield Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calabash, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tabor City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beaver, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Menomonee Falls, Wisconsin
- Croatia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dubrovnik
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varaždin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Denmark (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalborg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frederiksberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hillerød
- India (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bilāspur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Germán
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dos Hermanas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Cruz de Tenerife
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrevieja

REFERENCES:
- [Background] Grunberger G, Chang A, Garcia Soria G, Botros FT, Bsharat R, Milicevic Z. Monotherapy with the once-weekly GLP-1 analogue dulaglutide for 12 weeks in patients with Type 2 diabetes: dose-dependent effects on glycaemic control in a randomized, double-blind, placebo-controlled study. Diabet Med. 2012 Oct;29(10):1260-7. doi: 10.1111/j.1464-5491.2012.03745.x. PMID 22804250
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22804250

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.1 Milligrams (mg) LY2189265: LY2189265: 0.1 milligram (mg), subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
- 0.5 Milligrams (mg) LY2189265: LY2189265: 0.5 milligram (mg), subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
- 1.0 Milligrams (mg) LY2189265: LY2189265: 1.0 milligram (mg), subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
- 1.5 Milligrams (mg) LY2189265: LY2189265: 1.5 milligrams (mg), subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
- 3.0 Milligrams (mg) LY2189265: LY2189265: 3.0 milligram (mg), subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
- Placebo: Placebo: subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
Period: Overall Study
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | 3.0 Milligrams (mg) LY2189265 | Placebo
Started | 35 | 34 | 34 | 29 | 3 (3mg LY2189265 discont. Replaced with 1.5mg dose based on dose finding Study H9X-MC-GBCF; NCT00734474) | 32
Received at Least One Dose of Study Drug | 35 | 34 | 34 | 29 | 3 | 32
Completed | 33 | 31 | 34 | 25 | 0 | 29
Not Completed | 2 | 3 | 0 | 4 | 3 | 3
Not completed — Dose Discontinued per Sponsor Decision | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- 0.1 Milligrams (mg) LY2189265: LY2189265: 0.1 milligrams (mg), subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
- 0.5 Milligrams (mg) LY2189265: LY2189265: 0.5 milligrams (mg), subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
- 1.0 Milligrams (mg) LY2189265: LY2189265: 1.0 milligrams (mg), subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
- 1.5 Milligrams (mg) LY2189265: LY2189265: 1.5 milligrams (mg) subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
- Total: Total of all reporting groups
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | 3.0 Milligrams (mg) LY2189265 | Placebo | Total
Number analyzed (Participants) | 35 | 34 | 34 | 29 | 3 | 32 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.33 (9.15) | 56.91 (9.06) | 57.16 (8.76) | 57.45 (7.88) | 60.82 (7.15) | 55.03 (9.33) | 56.64 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 18 | 16 | 2 | 14 | 92
  Male | 11 | 16 | 16 | 13 | 1 | 18 | 75
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 0 | 0 | 0 | 3
  Asian | 4 | 5 | 5 | 4 | 0 | 5 | 23
  Black or African American | 1 | 1 | 0 | 1 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 29 | 28 | 26 | 24 | 2 | 25 | 134
  Multiple | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 13 | 11 | 3 | 17 | 75
  Mexico | 5 | 5 | 4 | 4 | 0 | 5 | 23
  Puerto Rico | 0 | 1 | 2 | 2 | 0 | 0 | 5
  Spain | 2 | 3 | 1 | 1 | 0 | 1 | 8
  Poland | 2 | 2 | 5 | 5 | 0 | 2 | 16
  Croatia | 4 | 2 | 2 | 3 | 0 | 3 | 14
  Russian Federation | 2 | 1 | 2 | 0 | 0 | 0 | 5
  India | 4 | 5 | 5 | 3 | 0 | 4 | 21
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meters (kg/m^2) | 32.92 (4.75) | 32.26 (5.39) | 32.22 (4.50) | 31.04 (4.29) | 35.38 (3.96) | 32.07 (5.23) | 32.20 (4.83)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 3.90 (3.19) | 3.72 (3.80) | 3.28 (2.54) | 4.62 (4.08) | 5.00 (3.04) | 3.91 (4.74) | 3.88 (3.68)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 87.08 (17.28) | 90.20 (21.34) | 86.89 (16.95) | 85.81 (18.63) | 100.90 (25.51) | 90.87 (18.94) | 88.43 (18.68)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 7.13 (0.55) | 7.18 (0.60) | 7.28 (0.66) | 7.25 (0.43) | 7.63 (0.15) | 7.36 (0.63) | 7.24 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: Least Squares (LS) means of change from baseline for glycosylated hemoglobin (HbA1c) were calculated using mixed model repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and baseline HbA1c as covariate.
Time Frame: Baseline, 12 weeks
Population: Participants who received at least one dose of study drug and have glycosylated hemoglobin (HbA1c) change from baseline data available. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Groups:
- 0.1 Milligrams (mg) LY2189265: LY2189265: 0.1 milligram (mg), subcutaneous (SC) injection, once weekly (QW), along with lifestyle measures for up to 12 weeks
- 0.5 Milligrams (mg) LY2189265: LY2189265 0.5 milligram (mg): subcutaneous (SC) injection, once weekly (QW), along with lifestyle measures for up to 12 weeks
- 1.0 Milligrams (mg) LY2189265: LY2189265 1.0 milligram (mg): subcutaneous (SC) injection, once weekly (QW), along with lifestyle measures for up to 12 weeks
- 1.5 Milligrams (mg) LY2189265: LY2189265 1.5 milligram (mg): subcutaneous (SC) injection, once weekly (QW), along with lifestyle measures for up to 12 weeks
- Placebo: Placebo: subcutaneous (SC) injection, once weekly (QW), along with lifestyle measures for up to 12 weeks
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 34 | 30 | 32 | 21 | 28
percentage of glycosylated hemoglobin | -0.37 (0.11) | -0.89 (0.12) | -1.03 (0.11) | -1.04 (0.13) | 0.01 (0.13)
Statistical Analysis 1: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265 vs Placebo; Test of log linear dose response with placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05
Statistical Analysis 2: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265; Test of log linear dose response without placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05
Statistical Analysis 3: Comparison: 0.1 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.069, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -0.37
Statistical Analysis 4: Comparison: 0.5 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -0.89
Statistical Analysis 5: Comparison: 1.0 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -1.04
Statistical Analysis 6: Comparison: 1.5 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -1.04

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and baseline glycosylated hemoglobin (HbA1c) as covariate.
Time Frame: Baseline, 4 weeks, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 35 | 34 | 34 | 26 | 29
percentage of glycosylated hemoglobin
  Week 4 (n=35, n=34, n=34, n=25, n=29) | -0.28 (0.09) | -0.51 (0.09) | -0.46 (0.08) | -0.53 (0.10) | -0.01 (0.10)
  Week 8 (n=35, n=30, n=33, n=24, n=28) | -0.33 (0.10) | -0.74 (0.10) | -0.78 (0.10) | -0.90 (0.12) | -0.00 (0.11)
Statistical Analysis 1: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265 vs Placebo; Test of log linear dose response with placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at Week 4. A priori threshold for statistical significance was p<0.05
Statistical Analysis 2: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265; Test of log linear dose response without placebo; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis — Treatment comparison at Week 4. A priori threshold for statistical significance was p<0.05
Statistical Analysis 3: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265 vs Placebo; Test of log linear dose response with placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at Week 8. A priori threshold for statistical significance was p<0.05
Statistical Analysis 4: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265; Test of log linear dose response without placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison at Week 8. A priori threshold for statistical significance was P<0.05

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: Fasting blood glucose is a test to determine how much glucose (sugar) is in a blood sample after an overnight fast. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and baseline fasting glucose as covariate.
Time Frame: Baseline, 12 weeks
Population: Participants who received at least one dose of study drug and have fasting blood glucose change from baseline data available. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Groups:
- 0.1 Milligrams (mg) LY2189265: LY2189265: 0.1 milligrams (mg), subcutaneous (SC) injection, once weekly (QW), along with lifestyle measures for up to 12 weeks
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 35 | 34 | 34 | 28 | 31
milligrams per deciliter (mg/dL) | -11.59 (4.09) | -30.31 (4.26) | -33.73 (4.18) | -37.49 (4.78) | -3.78 (4.44)
Statistical Analysis 1: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265 vs Placebo; Test of log linear dose response with placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05
Statistical Analysis 2: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265; Test of log linear dose response without placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05
Statistical Analysis 3: Comparison: 0.1 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.456, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -7.81
Statistical Analysis 4: Comparison: 0.5 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -26.53
Statistical Analysis 5: Comparison: 1.0 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -29.96
Statistical Analysis 6: Comparison: 1.5 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -33.71

4. Secondary Outcome: Percentage of Participants Who Achieve Glycosylated Hemoglobin (HbA1c) <7% or ≤6.5%
Description: Percentages of participants who achieved glycosylated hemoglobin (HbA1c) levels of <7.0% or ≤6.5% were compared across treatment arms using the Cochran-Armitage trend test.
Time Frame: 12 weeks
Population: Participants who received at least one dose of study drug and have HbA1c data available. Only pre-rescue measurements were used.
Measure: Number; unit: percentage of participants
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 35 | 34 | 34 | 29 | 32
percentage of participants
  HbA1c levels <7.0% (n=34, n=30, n=32, n=21, n=28) | 47.1 | 73.3 | 75.0 | 71.4 | 21.4
  HbA1c levels ≤6.5% (n=34, n=30, n=32, n=21, n=28) | 14.7 | 53.3 | 50.0 | 52.4 | 7.1
Statistical Analysis 1: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Armitage trend test — Treatment comparison of glycosylated hemoglobin (HbA1c) levels <7.0%; The Cochran-Armitage trend test included the placebo arm
Statistical Analysis 2: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Armitage trend test — Treatment comparison of glycosylated hemoglobin (HbA1c) levels ≤6.5%; The Cochran-Armitage trend test included the placebo arm

5. Secondary Outcome: Change From Baseline in Daily Mean Blood Glucose Values From the 7-point Self Monitored Blood Glucose (SMBG) Profiles
Description: Change from baseline in mean daily blood glucose values were measured with a 7-point self-monitored blood glucose (SMBG) profile over a 24-hour period in the 7-day period prior to each visit. The 7-point SMBG profile consisted of preprandial blood glucose measures before the morning, midday, and evening meals; blood glucose measures 2 hours after the start of the morning, midday, and evening meals; and the fasting blood glucose obtained the following morning. Mean at 12 weeks was assessed in all treatment groups. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and as covariate.
Time Frame: Baseline, 12 weeks
Population: Participants who received at least one dose of study drug and have blood glucose change from baseline data available. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 34 | 32 | 33 | 28 | 31
milligrams per deciliter (mg/dL) | -15.77 (4.74) | -32.21 (4.88) | -42.46 (4.68) | -44.79 (5.46) | -6.12 (5.05)
Statistical Analysis 1: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265 vs Placebo; Test of log linear dose response with placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05
Statistical Analysis 2: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265; Test of log linear dose response without placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05
Statistical Analysis 3: Comparison: 0.1 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.378, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -9.65
Statistical Analysis 4: Comparison: 0.5 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -26.09
Statistical Analysis 5: Comparison: 1.0 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -36.34
Statistical Analysis 6: Comparison: 1.5 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -38.67

6. Secondary Outcome: Change From Baseline in Beta-cell Function (HOMA2-%B)
Description: Change from baseline in beta (β)-cell function (HOMA2-%B) was assessed by using the homeostatic model assessment (HOMA) to quantify β-cell function. HOMA2-%B is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady state beta cell function (%B), as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. Least Squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and baseline HOMA2-%B as covariate.
Time Frame: Baseline, 12 weeks
Population: Participants who received at least one dose of study drug and have beta-cell function (HOMA2-%B) change from baseline data available. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2-%B
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 34 | 34 | 28 | 26 | 31
percentage of HOMA2-%B | 13.18 (6.76) | 31.66 (7.04) | 39.04 (7.64) | 29.29 (8.11) | -2.06 (7.44)
Statistical Analysis 1: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265 vs Placebo; Test of log linear dose response with placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05
Statistical Analysis 2: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265; Test of log linear dose response without placebo; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05

7. Secondary Outcome: Change From Baseline in Insulin Sensitivity (HOMA2-%S)
Description: Change from baseline in insulin sensitivity (HOMA2-%S) was assessed by using the homeostatic model assessment (HOMA) to quantify insulin sensitivity. HOMA2-%S is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady state insulin sensitivity (%S), as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. Least Squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and baseline HOMA2-%S as covariate.
Time Frame: Baseline, 12 weeks
Population: Participants who received at least one dose of study drug and have insulin sensitivity change from baseline data available. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2-%S
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 27 | 33 | 29 | 24 | 22
percentage of HOMA2-%S | -2.41 (6.62) | 6.10 (6.92) | -4.80 (7.44) | 12.98 (7.95) | 0.58 (7.34)
Statistical Analysis 1: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265 vs Placebo; Test of log linear dose response with placebo; Test type: Superiority or Other; p = 0.450, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05
Statistical Analysis 2: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265; Test of log linear dose response without placebo; Test type: Superiority or Other; p = 0.329, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05

8. Secondary Outcome: Change From Baseline in Electrocardiograms (ECGs) - Fridericia-corrected QT (QTcF) and PR Interval
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTc = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. The PR segment begins at the endpoint of the P wave and ends at the onset of the QRS complex. Least Squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and baseline measurement as covariate.
Time Frame: Baseline, 12 weeks
Population: Participants who received at least one dose of study drug and have Fridericia-corrected QT (QTcF) or PR interval change from baseline data available.
Measure: Least Squares Mean (Standard Error); unit: millisecond (msec)
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 32 | 31 | 34 | 25 | 29
millisecond (msec)
  Fridericia-corrected QT (QTcF) Interval | 1.34 (2.09) | -1.18 (2.11) | 4.56 (2.01) | -0.63 (2.33) | 0.70 (2.19)
  PR Interval | 3.22 (2.20) | 4.57 (2.23) | -0.55 (2.15) | 2.83 (2.46) | -0.89 (2.33)

9. Secondary Outcome: Change From Baseline in Electrocardiograms (ECGs) - Heart Rate
Description: Least Squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and baseline measurement as covariate.
Time Frame: Baseline, 12 weeks
Population: Participants who received at least one dose of study drug and have heart rate change from baseline data available.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 32 | 31 | 34 | 25 | 29
beats per minute (bpm) | 1.38 (1.48) | 1.16 (1.51) | 1.88 (1.44) | 4.18 (1.67) | 0.67 (1.58)

10. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Sitting pulse rate was measured. Least Squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and baseline measurement as covariate.
Time Frame: Baseline, 12 weeks
Population: Participants who received at least one dose of study drug and have pulse rate change from baseline data available.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 34 | 31 | 34 | 25 | 30
beats per minute (bpm) | 0.19 (1.44) | 0.25 (1.49) | 1.02 (1.43) | 1.34 (1.65) | 1.29 (1.54)

11. Secondary Outcome: Change From Baseline in Blood Pressure (BP)
Description: Sitting systolic blood pressure (SBP) and sitting diastolic blood pressure (DBP) were measured. Least Squares (LS) means of change were calculated using a mixed-effects model for repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and baseline measurement as covariate.
Time Frame: Baseline, 12 weeks
Population: Participants who received at least one dose of study drug and have blood pressure change from baseline data available.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 34 | 31 | 34 | 25 | 30
millimeters of mercury (mmHg)
  Sitting Systolic Blood Pressure | -2.21 (2.04) | 0.51 (2.12) | -2.57 (2.02) | 1.88 (2.33) | -0.68 (2.18)
  Sitting Diastolic Blood Pressure | -0.24 (1.21) | 0.59 (1.26) | 0.42 (1.20) | 1.56 (1.39) | 1.07 (1.30)

12. Secondary Outcome: Number of Participants With Self-reported Hypoglycemic Events
Description: Hypoglycemic events were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined an event during which typical symptoms of hypoglycemia were accompanied by a blood glucose level of ≤3.9 millimoles per liter [mmol/L]), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured blood glucose of ≤3.9 mmol/L), or nocturnal (defined as any hypoglycemic event that occurred between bedtime and breakfast with a measured blood glucose of ≤3.9 mmol/L). Participant reports of hypoglycemic events were collected at the beginning of each visit starting at Baseline. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 12 weeks
Population: Participants who received at least one dose of study drug and have self-reported hypoglycemic event data available. Only pre-rescue measurements were used.
Measure: Number; unit: participants
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 35 | 34 | 34 | 29 | 32
participants
  Documented Symptomatic | 0 | 2 | 2 | 3 | 0
  Asymptomatic | 1 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0
  Nocturnal | 1 | 2 | 1 | 2 | 0

13. Secondary Outcome: Rate of Self-reported Hypoglycemic Events
Description: Hypoglycemic events (HE) were classified as severe (defined as events requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined an event during which typical symptoms of hypoglycemia were accompanied by a blood glucose level of ≤3.9 millimoles per liter [mmol/L]), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured blood glucose of ≤3.9 mmol/L), or nocturnal (defined as any HE that occurred between bedtime and breakfast with a measured blood glucose of ≤3.9 mmol/L). Participant reports of HE were collected at the beginning of each visit starting at Baseline and the annualized rate was reported. Least Squares (LS) means rates were adjusted for pre-study therapy, country, and baseline body mass index. A summary of AEs regardless of causality is located in the Reported AEs module. Some model-adjusted LS means are less than 0 and may be interpreted as very low rates.
Time Frame: Baseline through 12 weeks
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Events per participant per year
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 35 | 34 | 34 | 29 | 32
Events per participant per year
  Documented Symptomatic Hypoglycemic Rate | -0.08 (0.72) | 0.25 (0.73) | 1.68 (0.73) | 0.61 (0.79) | -0.09 (0.75)
  Asymptomatic Hypoglycemic Rate | 0.19 (0.10) | -0.01 (0.10) | -0.01 (0.10) | 0.02 (0.11) | 0.01 (0.11)
  Severe Hypoglycemic Rate | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Nocturnal Hypoglycemic Rate | 0.20 (0.62) | 0.16 (0.64) | 1.21 (0.62) | 0.21 (0.71) | -0.08 (0.67)

14. Secondary Outcome: Treatment Emergent Adverse Events
Description: A treatment emergent adverse event is any untoward medical occurrence that either occurs or worsens at any time after the first injection of study drug following randomization and which does not necessarily have to have a causal relationship. The number of participants with one or more treatment emergent adverse event was reported. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 12 weeks
Population: Participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- 3.0 Milligrams (mg) LY2189265: LY2189265: 3.0 milligrams (mg) subcutaneous (SC) injection, once weekly (QW), along with life style changes for up to 12 weeks
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | 3.0 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 35 | 34 | 34 | 29 | 3 | 32
participants | 21 | 17 | 20 | 18 | 1 | 18

15. Secondary Outcome: Change From Baseline in Body Weight
Description: Least Squares (LS) means was calculated using a mixed-effects model for repeated measures (MMRM) with pre-study therapy, country, dose, visit, and dose-by-visit interaction as fixed effects and baseline measurement as covariate.
Time Frame: Baseline, 12 weeks
Population: Participants who received at least one dose of study drug and have body weight change from baseline data available.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 34 | 31 | 34 | 25 | 30
kilogram (kg) | -0.19 (0.42) | -0.34 (0.43) | -1.11 (0.42) | -1.49 (0.48) | -1.38 (0.45)
Statistical Analysis 1: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265 vs Placebo; Test of log linear dose response with placebo; Test type: Superiority or Other; p = 0.969, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05
Statistical Analysis 2: Comparison: 0.1 Milligrams (mg) LY2189265 vs 0.5 Milligrams (mg) LY2189265 vs 1.0 Milligrams (mg) LY2189265 vs 1.5 Milligrams (mg) LY2189265; Test of log linear dose response without placebo; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis — A priori threshold for statistical significance was p<0.05
Statistical Analysis 3: Comparison: 0.1 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.140, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = 1.19
Statistical Analysis 4: Comparison: 0.5 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.247, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = 1.04
Statistical Analysis 5: Comparison: 1.0 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.975, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = 0.27
Statistical Analysis 6: Comparison: 1.5 Milligrams (mg) LY2189265 vs Placebo; Test type: Superiority or Other; p = 1.00, Mixed Models Analysis — An adjustment for multiplicity was performed when comparing the individual doses to placebo using a Dunnett's test; Mean Difference (Final Values) = -0.11

16. Secondary Outcome: Antibody Production and Effects to LY2189265
Description: LY2189265 anti-drug antibodies (ADA) were assessed at baseline, 4 and 12 weeks, and at the safety follow-up visit 4 weeks after study drug discontinuation (16 weeks). The number of participants with initial postbaseline detection of treatment emergent (defined as a 4-fold increase in the ADA titer from baseline) LY2189265 ADA at each time point were summarized.
Time Frame: Baseline, 4 weeks, 12 weeks, 16 weeks
Population: Participants who received at least one dose of study drug with evaluable LY2189265 anti-drug antibodies (ADA) data.
Measure: Number; unit: participants
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | Placebo
Number analyzed (Participants) | 35 | 34 | 34 | 29 | 32
participants
  Week 4 | 0 | 0 | 1 | 0 | 0
  Week 12 | 0 | 0 | 0 | 0 | 0
  Week 16 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Collection and Evaluation of Plasma Levels (Pharmacokinetics [PK]) of LY2189265
Description: The population mean estimates and standard deviations were calculated for pharmacokinetic parameters (area under the concentration time curve (AUC) from zero to 168 hours). Evaluable PK concentrations from the 4 week, 8 week, and 12 week timepoints were combined and utilized in a population approach to determine the population mean estimate and standard deviation at steady-state.
Time Frame: 4 weeks, 8 weeks, 12 weeks
Population: Participants who received at least one dose of LY2189265 (0.1-3.0 milligrams [mg]) with evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | 3.0 Milligrams (mg) LY2189265
Number analyzed (Participants) | 27 | 31 | 34 | 27 | 2
nanograms*hour/milliliter (ng*h/mL) | 2294 (1503) | 6650 (4356) | 11671 (7645) | 16649 (10905) | 31538 (20657)

ADVERSE EVENTS:
Arm/Group | 0.1 Milligrams (mg) LY2189265 | 0.5 Milligrams (mg) LY2189265 | 1.0 Milligrams (mg) LY2189265 | 1.5 Milligrams (mg) LY2189265 | 3.0 Milligrams (mg) LY2189265 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/34 | 1/34 | 1/29 | 0/3 | 1/32
Other Adverse Events (participants affected / at risk) | 20/35 | 16/34 | 17/34 | 15/29 | 1/3 | 15/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.1 Milligrams (mg) LY2189265 (N=35) | 0.5 Milligrams (mg) LY2189265 (N=34) | 1.0 Milligrams (mg) LY2189265 (N=34) | 1.5 Milligrams (mg) LY2189265 (N=29) | 3.0 Milligrams (mg) LY2189265 (N=3) | Placebo (N=32)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 0.1 Milligrams (mg) LY2189265 (N=35) | 0.5 Milligrams (mg) LY2189265 (N=34) | 1.0 Milligrams (mg) LY2189265 (N=34) | 1.5 Milligrams (mg) LY2189265 (N=29) | 3.0 Milligrams (mg) LY2189265 (N=3) | Placebo (N=32)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (7) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hunger (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/24 (0) | 0/18 (0) | 0/18 (0) | 0/16 (0) | 0 (0) | 1/14 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days